CLINICAL TRIAL: NCT04492033
Title: A Phase 1b/2a Multi-center Study to Assess the Safety, Tolerability, Pharmacokinetics of CTX-009 (ABL001) in Combination With Irinotecan or Paclitaxel in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of CTX-009 (ABL001) in Combination With Irinotecan or Paclitaxel in Advanced or Metastatic Solid Tumor Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change of Development Plan
Sponsor: Handok Inc. (Industry)
Collaborators: Compass Therapeutics (Industry); ABL Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABL001-P1bC; CTX-009-001 (Other: Compass Therapeutics)
Record Dates: First submitted 2020-06-15; First posted 2020-07-30 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: P1b: Advanced Solid Tumors; P2: Biliary Tract Cancer
Keywords: VEGF; DLL4; Solid Tumors; Bispecific antibody; anti-angiogenic
MeSH Terms: interventions — asciminib; Paclitaxel; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CTX-009 (ABL001) and Paclitaxel (P1b) (Experimental)
  Interventions: Drug: CTX-009 (ABL001); Drug: Paclitaxel
- CTX-009 (ABL001) and Irinotecan (P1b) (Experimental): 1 cycle = 4weeks
  Interventions: Drug: CTX-009 (ABL001); Drug: Irinotecan
- CTX-009 (ABL001) and Paclitaxel (P2) (Experimental): 1 cycle = 4weeks
  Interventions: Drug: CTX-009 (ABL001); Drug: Paclitaxel

INTERVENTIONS:
Drug: CTX-009 (ABL001) — CTX-009 (ABL001) will be administered biweekly.
Drug: Paclitaxel — Paclitaxel will be administered weekly.
  Arms: CTX-009 (ABL001) and Paclitaxel (P1b); CTX-009 (ABL001) and Paclitaxel (P2)
Drug: Irinotecan — Irinotecan will be administered biweekly.
  Arms: CTX-009 (ABL001) and Irinotecan (P1b)

SUMMARY:
This study is a Phase 1b/2 multi-center study to assess the safety, tolerability, pharmacokinetics of CTX-009 (ABL001) in combination with Irinotecan or Paclitaxel in patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Phase 1b Study:

Indication of phase 1b study is the advanced or metastatic solid tumors (including, but not limited to, colorectal cancer, gastric cancer, and ovarian cancer).

Phase 2 Study:

Indication of phase 2 study is unresectable advanced, metastatic or recurrent biliary tract cancer (BTC) (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, gallbladder cancer, and ampullary carcinoma).

ELIGIBILITY:
Key Inclusion Criteria:

* P1b only: Patients with histologically or cytologically confirmed metastatic or unresectable advanced solid tumors
* P2 only: Patients with histologically or cytologically confirmed unresectable advanced, metastatic, or recurrent biliary tract cancers (including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, gallbladder cancer, ampullary carcinoma)
* P2 only: Patients who have shown disease progress or recurrence of disease after receiving first-line or second-line systemic chemotherapy, including treatment with gemcitabine in combination with a platinum agent
* Patients aged 19 years or older
* At least one lesion measurable defined by response evaluation criteria in solid tumors (RECIST) version 1.1.
* Life expectancy ≥ 12 weeks
* ECOG performance status 0 or 1
* Women of childbearing potential must have a negative pregnancy test outcome
* Patients must provide written informed consent to voluntary participation in this study

Key Exclusion Criteria:

* History of hypersensitivity reactions to any of the components of the investigational product or other drugs of the same class (humanized/human monoclonal antibody) and irinotecan or paclitaxel
* Less than 4 weeks have elapsed since a surgery
* History of cardiac illness: New York Heart Association (NYHA) class ≥ II congestive heart failure (CHF), uncontrolled hypertension, hypertension crisis, pulmonary hypertension, myocardial infarction, uncontrolled arrhythmia, unstable angina
* Persistent, clinically significant NCI-CTCAE v5.0 Grade ≥ 2 toxicities from the previous anticancer therapy
* Severe infections or major and unhealed injury (active ulcer, untreated fracture)
* Symptomatic or uncontrolled central nervous system (CNS) metastasis
* Pregnant or lactating women or patients planning to become pregnant during the study
* Participation in another clinical trial within 30 days prior to initiation of study treatment and received an investigational drug treatment
* Administration of antiplatelets or anticoagulants within 2 weeks prior to screening
* Requiring continuous treatment with systemic NSAIDs or systemic corticosteroids
* HIV or other severe diseases that warrant the exclusion from this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
P1b: Proportion of subjects with Dose-Limiting Toxicity (DLT) | From Day 1 until disease progression or Day 28, whichever came first
  Number of subjects who experience DLT events during 28 days after first administration of CTX-009 (ABL001) and Irinotecan/Paclitaxel, divided by the number of DLT-evaluable subjects
P2: Objective response rate (ORR) of CTX-009 (ABL001) in combination with paclitaxel in patients with BTC | Up to approximately 24 months
  The proportion of subjects whose best overall response (BOR) is assessed to be complete response (CR) or partial response (PR) as per Independent Radiology Center's review

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 24 months
  Severity of AEs will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Pharmacokinetics (PK) of CTX-009 (ABL001) | Up to approximately 24 months
  Serum concentrations of CTX-009 (ABL001) will be collected and analyzed to evaluate the PK of CTX-009 (ABL001)
Objective response rate (ORR) | Up to approximately 24 months
  Proportion of subject with best overall response of complete response (CR) or partial response (PR) as per investigator's review
Disease control rate (DCR) | Up to approximately 24 months
  Proportion of subjects with a best overall response of complete response (CR), partial response (PR) or stable disease (SD)
Time to treatment failure (TTF) | Up to approximately 24 months
  Time interval from 1st administration of CTX-009 (ABL001) to the time of disease progression or discontinuation of CTX-009 (ABL001) due to whatever reason, whichever comes first
Duration of response (DOR) | Up to approximately 24 months
  Time interval from first occurrence of a documented objective response to the time of disease progression
Progression-free survival (PFS) | Up to approximately 24 months
  The time from the initiation of treatment to the first radiologic assessment that confirms progression of tumor or to death
P2: Survival rate | 6 months and 12 months
  The proportion of subjects who have survived at 6 months and 12 months from the initiation of treatment
P2: Overall survival (OS) | Up to approximately 24 months
  Time from the initiation of treatment to death

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided